CLINICAL TRIAL: NCT06462313
Title: Director, Head of Anesthesiology and Critical Care, Principal Investigator, Professor
Brief Title: Dobutamine for Management of Surgical Patients With Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Ningbo No. 1 Hospital (Other); Lishui Country People's Hospital (Other); The Central Hospital of Lishui City (Other); Zhejiang Provincial Tongde Hospital (Other); Ningbo No.2 Hospital (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Zunyi Medical College (Other); The Second Hospital of Hebei Medical University (Other); Affiliated Hospital of Jiaxing University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Huaibei Peolple's Hospital (Unknown); Anqing People's Hospital of Anhui Medical University (Unknown); The Second Hospital University of South China (Other); The First Affiliated Hospital of University of South China (Other); Wenzhou people's hospitalï¼Œzhejiang province,China (Unknown); People's Hospital of Xinjiang Uygur Autonomous Region (Other); The First Clinical College of Harbin University (Unknown); The First Affiliated Hospital of Shihezi University Medical College (Unknown); Weifang People's Hospital (Other); Tianjin Medical University General Hospital (Other); Central Hospital of Heng Yang (Unknown); First Affiliated Hospital of Shenzhen University (Unknown); Henan Provincial People's Hospital (Other); Southwest Hospital, China (Other); The First People's Hospital of Zunyi (Other); Affiliated Hospital of Guangdong Medical University (Other); Union hospital of Fujian Medical University (Other); Bijie Hospital of Zhejiang Provincial People's Hospital (Unknown); Red Cross Hospital, Hangzhou, China (Other); Weihai Municipal Hospital (Other); The First Affiliated Hospital of Soochow University (Other); Zhejiang Cancer Hospital (Other); Renmin Hospital of Wuhan University (Other); Wuhan Third Hospital (Other); Tongji Hospital (Other); Zhujiang Hospital (Other); Fuyang Hospital of Anhui Medical University (Unknown); The Hospital of Suixi County (Unknown); Fujian Provincial Hospital (Other); Guizhou Provincial People's Hospital (Other); Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, xiangming fang, professor, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dobutamine
Record Dates: First submitted 2024-05-23; First posted 2024-06-17 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Patients With Septic Shock; Surgical Patients; General Anesthesia
MeSH Terms: interventions — Dobutamine; Norepinephrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dobutamine, norepinephrine (Experimental): Patients will be initiated on Dobutamine at 5 mcg/kg/min while continuous infusion of norepinephrine titrated to maintain a mean arterial pressure at 65mmHg or more
  Interventions: Drug: Dobutamine; Drug: Norepinephrine
- Norepinephrine (Other): Norepinephrine was titrated to maintain a mean arterial pressure at 65mmHg or more
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Dobutamine — Patients with septic shock in Dobutamine group will be initiated on Dobutamine at 5 mcg/kg/min when electrocardiogram, invasive blood pressure, and oxygen saturation were monitored.
  Arms: Dobutamine, norepinephrine
Drug: Norepinephrine — Norepinephrine was titrated to maintain a mean arterial pressure at 65mmHg or more in both groups.

SUMMARY:
Septic shock is the last and most severe stage of sepsis and is defined by extremely low blood pressure, despite lots of intravenous fluids. The incidence of septic shock related cardiomyopathy was 10% to 70%. Besides, general anesthesia will inhibit the sympathetic nervous system, reduce myocardial contractility and aggravate cardiac dysfunction. No randomized controlled trials have yet explore the effects of dobutamine on clinical outcomes for patients with septic shock undergoing surgery under general anesthesia.

DETAILED DESCRIPTION:
Sepsis, defined as life-threatening organ dysfunction, is caused by a dysregulated host response to infection, which 30-day mortality rate is about 24.4%. Septic shock is the last and most severe stage of sepsis and is defined by extremely low blood pressure, despite lots of intravenous fluids.

Surgical patients with septic shock are not rare. The incidence of septic shock related cardiomyopathy was 10% to 70%. Besides, general anesthesia will inhibit the sympathetic nervous system, reduce myocardial contractility and aggravate cardiac dysfunction, furthermore exacerbate hemodynamic instability, and then increase the incidence of AKI and patient mortality. Therefore, to improve cardiac function in patients with septic shock who received general anesthesia is the key to save patients life and improve prognosis.

The latest international guidelines for the treatment of septic shock recommend - in patients with septic shock combined with cardiac dysfunction, treatment with norepinephrine in combination with dobutamine is recommended if inadequate tissue perfusion persists after adequate fluid resuscitation and maintenance of blood pressure, but the level of evidence is weak.

Dobutamine acts on β-adrenergic receptors, which can improve tissue perfusion, and small doses of 2.5-5ug/kg/min can increase myocardial contractility and improve cardiac function in patients without increasing heart rate. Previous study has demonstrated that the combined use of norepinephrine and dobutamine can elevate left ventricular ejection fraction, cardiac index, improve tissue perfusion, and reduce mortality in patients with septic shock. No randomized controlled trials have yet explore the effects of dobutamine on clinical outcomes for patients with septic shock undergoing surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with 18 years or older
2. Sugery patients with septic shock and the duration of opration is more than 1 hour

Exclusion Criteria:

1. Pregnancy;
2. Long-term intakeβ-receptor blocker;
3. patietns with dobutamine used within 72h before enrollment;
4. Patients use Recombinant Human Brain Natriuretic Peptide(rhBNP), Levosimendan and Epinephrine within 72h before enrollment;
5. Patients with hyperthyroidism;
6. Allergy or known sensitivity to catecholamines（norepinephrine, dobutamine etc.）and genera anesthetics.
7. Patients and guardians refused to participate in this intervention clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Incidence of acute kidney injury after surgery | within 1 week after surgery
  Incidence of acute kidney injury after surgery
Sequential Organ Failure Assessment (SOFA) score | Day 1 Day 3 and Day 7 in ICU after surgery
  Sequential Organ Failure Assessment (SOFA) score, ranges from 0 to 24, with 24 being the worst
Mortality | in hospital and Day 28 and Day 90 after the surgery
  Mortality

SECONDARY OUTCOMES:
Lactate level measurement | before surgery (0 hour), 1hour after begining of surgery and at the end of surgey
  Lactate level measurement
capillary filling time | before surgery (0 hour), 1hour after begining of surgery and at the end of surgey
  capillary filling time
Central venous oxygen saturation (ScvO2) | before surgery (0 hour), 1hour after begining of surgery and at the end of surgey
  Central venous oxygen saturation (ScvO2)
Urine volume | 1hour after begining of surgery and at the end of surgey
  Urine volume
Duration of norepinephrine intraoperatively | intraoperatively
  Duration of norepinephrine intraoperatively
Cumulative dose of norepinephrine intraoperatively | intraoperatively
  Cumulative dose of norepinephrine intraoperatively
Incidence of intraoperative arrythmia Incidence of intraoperative arrythmia | intraoperatively
  Incidence of intraoperative arrythmia
Postoperative complication | through study completion, an average of 1 year
  Postoperative complication
Length of hospital stay after sugery | through study completion, an average of 1 year
  Length of hospital stay after sugery
ICU-free days with 28 days postoperatively | 28 days postoperatively
  ICU-free days with 28 days postoperatively
Duration of mechanical ventilation in ICU | through study completion, an average of 1 year
  Duration of mechanical ventilation in ICU
Renal replacement therapy | through study completion, an average of 1 year
  Renal replacement therapy within the first 7 days after the surgery
Duration of renal replacement therapy | through study completion, an average of 1 year
  Duration of renal replacement therapy
ICU-Mortality | through study completion, an average of 1 year
  ICU-Mortality
In-hosipital Mortality | through study completion, an average of 1 year
  In-hosipital Mortality
Hospitalization costs | through study completion, an average of 1 year
  Hospitalization costs

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol
Supporting Information: Study Protocol
Time Frame: after finishing the study
Access Criteria: The protocol is available from the investigator on reasonable request.

REFERENCES:
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Bauer M, Gerlach H, Vogelmann T, Preissing F, Stiefel J, Adam D. Mortality in sepsis and septic shock in Europe, North America and Australia between 2009 and 2019- results from a systematic review and meta-analysis. Crit Care. 2020 May 19;24(1):239. doi: 10.1186/s13054-020-02950-2. PMID 32430052
- [Background] Singbartl K, Kellum JA. AKI in the ICU: definition, epidemiology, risk stratification, and outcomes. Kidney Int. 2012 May;81(9):819-25. doi: 10.1038/ki.2011.339. Epub 2011 Oct 5. PMID 21975865
- [Background] Liu J, Xie H, Ye Z, Li F, Wang L. Rates, predictors, and mortality of sepsis-associated acute kidney injury: a systematic review and meta-analysis. BMC Nephrol. 2020 Jul 31;21(1):318. doi: 10.1186/s12882-020-01974-8. PMID 32736541
- [Background] Uchino S, Kellum JA, Bellomo R, Doig GS, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Ronco C; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Acute renal failure in critically ill patients: a multinational, multicenter study. JAMA. 2005 Aug 17;294(7):813-8. doi: 10.1001/jama.294.7.813. PMID 16106006
- [Background] Yang HS, Song BG, Kim JY, Kim SN, Kim TY. Impact of propofol anesthesia induction on cardiac function in low-risk patients as measured by intraoperative Doppler tissue imaging. J Am Soc Echocardiogr. 2013 Jul;26(7):727-35. doi: 10.1016/j.echo.2013.03.016. Epub 2013 Apr 24. PMID 23622885
- [Background] Green DW. Cardiac output decrease and propofol: what is the mechanism? Br J Anaesth. 2015 Jan;114(1):163-4. doi: 10.1093/bja/aeu424. No abstract available. PMID 25500400
- [Background] Rudiger A, Singer M. Mechanisms of sepsis-induced cardiac dysfunction. Crit Care Med. 2007 Jun;35(6):1599-608. doi: 10.1097/01.CCM.0000266683.64081.02. PMID 17452940
- [Background] Zhu Y, Yin H, Zhang R, Ye X, Wei J. The effect of dobutamine in sepsis: a propensity score matched analysis. BMC Infect Dis. 2021 Nov 11;21(1):1151. doi: 10.1186/s12879-021-06852-8. PMID 34758739